CLINICAL TRIAL: NCT02590367
Title: Huo JieGe, Doctor of Medicine,Professor of Medicine,Professor of Medical Science.
Brief Title: Estimate the Efficacy of HD6610 Granule for Oxaliplatin-induced Peripheral Neuropathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, JieGe Huo, Huo JieGe, Doctor of Medicine,Professor of Medicine,Professor of Medical Science., Jiangsu Province Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JiangsuPHTCM
Record Dates: First submitted 2015-09-14; First posted 2015-10-29 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Peripheral Neuropathy
Keywords: oxaliplatin-induced peripheral neuropathy; HD6610 granule; colorectal cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Colorectal Neoplasms | interventions — Folfox protocol; XELOX

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOLFOX regimen&HD6610 Granule (Experimental): Patients in this group will be given conventional oxaliplatin based chemotherapy recommended by treatment guidelines for colorectal cancer, and the HD6610 Granule will be given 2 times a day.
  Interventions: Drug: FOLFOX regimen; Drug: HD6610 Granule
- FOLFOX regimen&HD6610 Granule placebo (Placebo Comparator): Patients in this group will be given conventional oxaliplatin based chemotherapy recommended by treatment guidelines for colorectal cancer, and the placebo HD6610 Granule
  Interventions: Drug: FOLFOX regimen; Drug: HD6610 Granule placebo

INTERVENTIONS:
Drug: FOLFOX regimen — FOLFOX regimens are combination therapy of oxaliplatin (85 mg/m^2) administered as a 2-hour infusion on Day 1; leucovorin (400 mg/m^2) administered as a 2-hour infusion on Day 1; followed by a loading dose of 5-fluorouracil (5-FU; 400 mg/m^2) IV bolus administered over approximately 2 to 4 minutes on Day 1, then 5- FU (different dose like FOLFOX4/FOLFOX6) via ambulatory pump administered for a period of 46 to 48 hours.
  XELOX is a combination therapy of Oxaliplatin 130mg/ m^2 d1 Intravenous infusion, every 3 weeks. and Capecitabine 1000mg/m^2 bid, days 1-14, every 3 weeks.
  Other Names: XELOX
Drug: HD6610 Granule — the HD6610 Granule will be given 2 times a day.
  Arms: FOLFOX regimen&HD6610 Granule
Drug: HD6610 Granule placebo — the HD6610 Granule placebo will be given 2 times a day.
  Arms: FOLFOX regimen&HD6610 Granule placebo

SUMMARY:
The purpose of this study is to estimate the usefulness and safety of HD6610 granule for oxaliplatin-induced peripheral neuropathy. The investigators examined the efficacy and safety of the treatment algorithm for 64 patients with colorectal cancer by evaluating the side effects and degree of improvement of subjective symptoms.

DETAILED DESCRIPTION:
Oxaliplatin is the third generation platinum-based cytotoxic agent, widely used in colorectal cancer, in metastatic disease and in the adjuvant setting . Moreover, oxaliplatin is being used as an alternative option to cisplatin in various cancers, such as ovarian, gastric. Oxaliplatin-induced peripheral neuropathy is characterised by acute and transient cold hyperaesthesia in the hours and days following oxaliplatin infusion (>90% of patients), but also by retarded chronic neuropathy due to the repetition of chemotherapy cycles (30-50% of patients). Oxaliplatin-induced peripheral neuropathy impairs the health-related quality of life (HRQOL) of patients and no preventive or curative strategies have as yet proven effective so far. Animal experiment show that HD6610 granule can relieve mouse's peripheral neuropathy induced by oxaliplatin. In clinical practice, the investigators also find that HD6610 granule can relieve patient's oxaliplatin-induced peripheral neuropathy in the treatment of chemotherapy. So the investigators design this randomized, parallel-group, double-blind, placebo-controlled, multicenter clinical study to estimate the efficacy and safety of HD6610 granule for oxaliplatin-induced peripheral neuropathy in colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. All cases have been diagnosed with colorectal cancer by pathology;
2. Patients who received no chemotherapy before should receive oxaliplatin-based chemotherapy(FOLFOX4,FOLFOX6,XELOX) ;
3. Patients of 18-70 years old have no serious heart,liver,kidney and hematopoietic disfunction,life expectancy of over 3 months and KPS more than 60;
4. Patients with no positive sign in neurological examination,and no drug allergy history or diabetes;
5. Volunteered to participate and signed informed consent,patients can not receive radiotherapy,acupuncture and moxibustion or other treatment during the experiment.

Exclusion Criteria:

1. Not accordant with the inclusion criteria;
2. Patients who have used herbal within 4 weeks before registration;
3. Patients who have serious heart,liver,kidney and hematopoietic disfunction;
4. Patients of central nervous system disease;
5. Patients of cervical spondylopathy,lumbar disc protrusion,diabetes and uremia which can potentially cause peripheral neuropathy;
6. Nerve compression caused by tumor metastasis or peripheral neuropathy caused by electrolyte disturbances,diabetes,alcohol disease and other disorder;
7. Long-time using of thiazide diuretic and foxglove;
8. Patients of poisoning,infection and radiotherapy which induced peripheral neuropathy or receiving medicine which can cause peripheral neuropathy;
9. Patients who can hardly take Chinese Medicine with severe diarrhea,vomiting or intestinal obstruction ;
10. Uncontrolled psychosis;
11. Women of pregnancy ,preparing pregnant, or lactation;
12. Alcohol and drug abuse;
13. Allergic constitution or allergy to experiment drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The number of patients with different degree of peripheral nerve toxicity. | Through study completion, an average of 1 year.

SECONDARY OUTCOMES:
EORTC（European Organization for Research and Treatment of Cancer） quality of life score | Through study completion, an average of 1 year.
KPS（ Karnofsky Performance Status Scale） score | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Huo JieGe, M.D., Study Director — Jiangsu Province Hospital of Traditional Chinese Medicine
Locations (1):
- Jiangsu Province Hospital of Integrated Chinese and Western Medicine, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Balayssac D, Ferrier J, Pereira B, Gillet B, Petorin C, Vein J, Libert F, Eschalier A, Pezet D. Prevention of oxaliplatin-induced peripheral neuropathy by a polyamine-reduced diet-NEUROXAPOL: protocol of a prospective, randomised, controlled, single-blind and monocentric trial. BMJ Open. 2015 Apr 1;5(4):e007479. doi: 10.1136/bmjopen-2014-007479. PMID 25833669